CLINICAL TRIAL: NCT01178801
Title: Sharable Knowledge Mining Platform for Clinical Data Extraction, and Medical Knowledge and Mining Services Sharing
Brief Title: Sharable Knowledge Mining Platform
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Feipei Lai/Professor & Director, National Taiwan University,Graduate Institute of Biomedical Electronics and Bioinformatics
Other Study IDs: 201002032R
Record Dates: First submitted 2010-05-30; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-07

CONDITIONS: Liver Cancer
Keywords: liver cancer; data mining; knowledge discovering; The clinical data of the patients with liver cancer.
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- liver cancer: Clinical data of patients with liver cancer

SUMMARY:
As a result of increasing adoption of health information systems in hospitals, more and more health records can be gathered and accumulated in the healthcare data repository. For this reason, the opportunity of analyzing and mining the healthcare data for quality improvement is increasing and becoming more and more important.

The purpose of the project is to gather the clinical data relevant to liver cancer, and adopt the knowledge discovery and mining modules in information technology (IT) for analyzing and discovering the knowledge from the gathered clinical data.

We can analyze the gathered clinical data for comparing the outcomes of different treatment strategies, finding out new diagnosis and staging criteria and factors, and other hidden knowledge included in the clinical data.

Afterwards, the discovered results and the mining algorithms can be shared though the sharable knowledge mining platform provided by our project.

ELIGIBILITY:
Inclusion Criteria:

* Clinical data of patients with liver cancer. (ICD9 Code is 155.0)
* Males and females

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with liver cancer. (ICD9 Code is 155.0)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
the relationship between the clinical data and the decision of treatment strategies | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Feipei Lai, Ph.D., Study Chair — National Taiwan University,Graduate Institute of Biomedical Electronics
Locations (1):
- National Taiwan University, Taipei, Taiwan